CLINICAL TRIAL: NCT01470313
Title: A Randomized, Subject And Investigator-Blinded (Sponsor-Open), Placebo-Controlled Study To Evaluate The Safety, Tolerability, And Preliminary Efficacy Of Multiple Ascending Doses Of PD- 0360324 In Subjects With Active Cutaneous Lupus Erythematosus (CLE)
Brief Title: A Multiple Dose Study Of PD-0360324 In Patients With Active Cutaneous Lupus Erythematosus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A6261008
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: Safety and tolerability; cutaneous lupus erythematosus; efficacy
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PD-0360324 (Experimental)
  Interventions: Drug: PD-0360324
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PD-0360324 — Subjects will receive PD-0360324 intravenously in 3 different cohorts. The cohorts will be evaluated in ascending fashion. The doses planned are 100 mg every other week for 3 months, 150 mg every other week for 3 months, and 200 mg every 4 weeks for 3 months.
  Arms: PD-0360324
Drug: Placebo — Placebo is normal saline. The timing of placebo administration will depend of the dosing frequency of the cohort (either every other week for 3 months or every 4 weeks for 3 months).
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and tolerability of multiple intravenously administered doses of PD-0360324 in patients with cutaneous lupus erythematosus. Changes in disease activity will also be evaluated.

DETAILED DESCRIPTION:
The trial was terminated prematurely on Oct 15, 2013 due to a business decision. The decision to terminate the trial was not based on any clinical safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects between the ages of 21 to 70 who have a clinical diagnosis of either discoid cutaneous lupus erythematosus or subacute cutaneous lupus erythematosus with or without systemic lupus erythematosus prior to screening that has been confirmed by evaluation of skin biopsy sample.
* Active disease at both screening and baseline (Day 1) defined by a CLASI score of greater than or equal to 10.
* Intolerance to antimalarial therapy or more than 3 months of antimalarial therapy with disease activity.

Exclusion Criteria:

* Use of greater than or equal to 20 mg or prednisone (or equivalent) within 3 months of Day 1.
* Signs or symptoms or relevant history of a viral, bacterial, fungal, and parasitic infection, or recent history of repeated infections
* Subjects with evidence of past or active tuberculosis
* Pregnant, planning to get pregnant, and/or lactating females or males planning to father a child within time period of the study or subsequent exclusionary period.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PD- 0360324 will be assessed by physical examinations, adverse event and infection monitoring, 12 lead ECGs, vital sign, and clinical safety laboratory measurements. | 16 Weeks

SECONDARY OUTCOMES:
Efficacy of PD-0360324 based upon reduction of severity of symptoms as measured using the activity score of the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) | 12 Weeks
Measure changes in systemic features using the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | 12 Weeks
Measure changes in biomarkers | 12 weeks
Assess health outcomes measures | 12 Weeks
Evaluate the Pharmacokinetics of PD-0360324 | 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (16):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Oxford, Alabama
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Orange Park, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Fort Gratiot, Michigan
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Ducansville, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Rapid City, South Dakota
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Clarksburg, West Virginia
- Pfizer Investigational Site, Markham, Ontario, Canada
- Pfizer Investigational Site, Chisinau, Moldova

REFERENCES:
- [Derived] Masek-Hammerman K, Peeva E, Ahmad A, Menon S, Afsharvand M, Peng Qu R, Cheng JB, Syed J, Zhan Y, O'Neil SP, Pleasic-Williams S, Cox LA, Beidler D. Monoclonal antibody against macrophage colony-stimulating factor suppresses circulating monocytes and tissue macrophage function but does not alter cell infiltration/activation in cutaneous lesions or clinical outcomes in patients with cutaneous lupus erythematosus. Clin Exp Immunol. 2016 Feb;183(2):258-70. doi: 10.1111/cei.12705. Epub 2015 Nov 9. PMID 26376111
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6261008&StudyName=A%20Multiple%20Dose%20Study%20Of%20PD-0360324%20In%20Patients%20With%20Active%20Cutaneous%20Lupus%20Erythematosus